CLINICAL TRIAL: NCT06652737
Title: Age De-escalation Clinical Trial to Evaluate the Safety, Tolerability and Immunogenicity of a Late Liver Stage-arresting, Replication-competent Plasmodium Falciparum Sporozoite Vaccine (Sanaria® PfSPZ-LARC2 Vaccine) Administered by Direct Venous Inoculation to Malaria-exposed Adults and Children in Burkina Faso
Brief Title: Age De-escalation Safety Trial of PfSPZ-LARC2 Vaccine in Burkina Faso
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sanaria Inc. (Industry)
Collaborators: University of Maryland, Baltimore (Other); Groupe de Recherche Action en Sante (Other); Seattle Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: BFSPZL1
Record Dates: First submitted 2024-10-18; First posted 2024-10-22 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Malaria Falciparum; Malaria Infection
Keywords: malaria; PfSPZ-LARC2 Vaccine; falciparum
MeSH Terms: conditions — Malaria, Falciparum; Malaria | interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: The first study groups will assess 2 doses of vaccine, the target dose (2x10e5 PfSPZ) and a "maximize-the-chances-of-breakthrough" 2-fold higher dose (4x10e5 PfSPZ). These 2 doses will be assessed in adults (cohort 1). After SMC review of safety data from these two groups, the trial will proceed to older children (cohort 2) and then younger children (cohort 3).
  Each age strata will receive a single immunization, except for group 1 (adults), which will receive three immunizations on days 1, 29 and 57. The reason for a single immunization is that the chance of breakthrough will diminish after the first dose due to the induction of immunity - thus, repeat doses are not expected to contribute more information. However, with group 1, second and third immunizations will be administered to be sure that there is no increase in reactogenicity with repeated dosing and also to address the hypothetical concern that the attenuation of second and third doses is different from what we expect
Who Masked: Participant, Care Provider, Investigator
Masking Description: parasitology teams laboratory teams clinical teams
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (10):
- Cohort 1: Group 1a Adult 2x10e5 PfSPZ-LARC2 Vaccine (Experimental): 20-50-year-olds: 10 participants receive 3 injections of 2.0x10e5 PfSPZ-LARC2 Vaccine
  Interventions: Biological: PfSPZ-LARC2 Vaccine
- Cohort 1: Group 1b Adult Normal Saline (Placebo Comparator): 20-50-year-olds: 5 participants receive 3 injections of normal saline
  Interventions: Biological: Normal Saline (Placebo)
- Cohort 1: Group 2a Adult 4x10e5 PfSPZ-LARC2 Vaccine (Experimental): 20-50-year-olds: 10 participants receive single injection of 4.0x10e5 PfSPZ-LARC2 Vaccine
  Interventions: Biological: PfSPZ-LARC2 Vaccine
- Cohort 2: Group 3a 11-17year old 2x10e5 PfSPZ-LARC2 Vaccine (Experimental): 11-17-year-olds: 10 participants receive single injection of 2.0x10e5 PfSPZ-LARC2 Vaccine
  Interventions: Biological: PfSPZ-LARC2 Vaccine
- Cohort 2: Group 3b 11-17 year-olds Normal Saline (Placebo Comparator): 11-17-year-olds: 5 participants receive single injection of Normal Saline
  Interventions: Biological: Normal Saline (Placebo)
- Cohort 2: Group 4a 6-10-year old 2x10e5 PfSPZ-LARC2 Vaccine (Experimental): 6-10-year-olds: 10 participants receive single injection of 2.0x10e5 PfSPZ-LARC2 Vaccine
  Interventions: Biological: PfSPZ-LARC2 Vaccine
- Cohort 2: Group 4b 6-10-year old Normal Saline (Placebo Comparator): 6-10-year-olds: 5 participants receive single injection of Normal Saline
  Interventions: Biological: Normal Saline (Placebo)
- Cohort 3: Group 5a 1-5-year old 2x10e5 PfSPZ-LARC2 Vaccine (Experimental): 1-5-year-olds: 10 participants receive one injection of 2.0x10e5 PfSPZ-LARC2 Vaccine
  Interventions: Biological: PfSPZ-LARC2 Vaccine
- Cohort 3: Group 5b 1-5-year old Normal Saline (Placebo Comparator): 1-5-year-olds: 5 participants receive one injection of Normal Saline
  Interventions: Biological: Normal Saline (Placebo)
- Cohort 1: Group 2b: Adults Normal Saline (Placebo Comparator): 20-50 year olds: 5 participants receive single injection of Normal Saline
  Interventions: Biological: Normal Saline (Placebo)

INTERVENTIONS:
Biological: PfSPZ-LARC2 Vaccine — The PfSPZ comprising PfSPZ-LARC2 Vaccine contain a double genetic deletion, of the Mei2 and LINUP genes, and undergo developmental arrest in the late liver stages without releasing merozoites into the blood stream (no blood stage parasites are produced)
  Arms: Cohort 1: Group 1a Adult 2x10e5 PfSPZ-LARC2 Vaccine; Cohort 1: Group 2a Adult 4x10e5 PfSPZ-LARC2 Vaccine; Cohort 2: Group 3a 11-17year old 2x10e5 PfSPZ-LARC2 Vaccine; Cohort 2: Group 4a 6-10-year old 2x10e5 PfSPZ-LARC2 Vaccine; Cohort 3: Group 5a 1-5-year old 2x10e5 PfSPZ-LARC2 Vaccine
Biological: Normal Saline (Placebo) — Normal Saline Placebo
  Arms: Cohort 1: Group 1b Adult Normal Saline; Cohort 1: Group 2b: Adults Normal Saline; Cohort 2: Group 3b 11-17 year-olds Normal Saline; Cohort 2: Group 4b 6-10-year old Normal Saline; Cohort 3: Group 5b 1-5-year old Normal Saline

SUMMARY:
This is a first-in-humans randomized, double-blind, placebo-controlled, age de-escalation Phase 1 trial of Plasmodium falciparum (Pf) late liver stage-arresting replication-competent (LARC) sporozoite (SPZ) malaria vaccine (Sanaria® PfSPZ-LARC2 Vaccine) administered to healthy, malaria-exposed adults and children by direct venous inoculation (DVI) to determine safety, tolerability, and immunogenicity. The PfSPZ comprising PfSPZ-LARC2 Vaccine contain a double gene deletion, of the Mei2 and LINUP genes. As a result, they undergo developmental arrest in the late liver stages without releasing merozoites into the blood stream (no blood stage parasites are produced, either asexual or sexual). Because Pf parasites with the LARC phenotype replicate in the liver before disintegrating, they amplify and diversify parasite protein expression and are expected to be a potent immunogen to induce anti-malarial immunity, equaling or exceeding the potency and efficacy of the replication-competent chemo-attenuated Sanaria® PfSPZ-CVac (chloroquine). Because the parasites are intrinsically attenuated, they are also expected to be safe and well tolerated, similar to radiation-attenuated Sanaria® PfSPZ Vaccine and to the single-gene(Mei2)-deleted GA2 parasites (also LARC phenotype) tested at the Leiden University Medical Center (LUMC), which, like PfSPZ-LARC2 Vaccine, disintegrate after replicating in the liver. PfSPZ-LARC2 Vaccine thus avoids the safety concerns associated with PfSPZ-CVac, which uses fully infectious, non-attenuated parasites to achieve replication and depends on co-administered chloroquine for attenuation. In summary, the genetically attenuated PfSPZ-LARC2 Vaccine should combine the best-in-class immunogenic potency and protective efficacy of PfSPZ-CVac (chloroquine) with the excellent safety and tolerability of intrinsically attenuated PfSPZ Vaccine and GA2 vaccine.

This trial is designed to test the hypotheses that:

1. The vaccine is safe and well tolerated in each age group.
2. The true rate of breakthrough blood stage infection (or other concerning adverse events) is less than about 5%, with an 95% confidence level (this will be the level of confidence that there are no breakthroughs if no breakthroughs occur in the 50 participants receiving PfSPZ-LARC2 Vaccine).

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, single-center Phase 1 clinical trial. The dose of PfSPZ to be tested in all age groups is 2.0x10e5, the same as the dose used in an NIH study of PfSPZ-CVac (chloroquine) which resulted in 100% vaccine efficacy against a heterologous controlled human malaria infection (CHMI) conducted 12 weeks after immunization]. 100% heterologous protection at 12 weeks represents the best protection ever recorded for a malaria vaccine. The selected dose, 2.0x10e5 PfSPZ, is roughly similar to the dose used in the GA2 study at LUMC. In one of the two adult groups, however, the 10 participants receiving vaccine will be administered a two-fold higher dose - 4.0x10e5 PfSPZ - to assess the risk of breakthrough more stringently in a malaria-experienced adult population at low risk for serious complications of malaria infection. If this high dose of PfSPZ does not lead to breakthrough in adults, it is unlikely that a 2-fold lower dose will lead to breakthrough in children.

There will be three cohorts of participants initiated in staggered fashion. These consist of 2 groups of adults in cohort 1 (receiving, respectively, 2.0x10e5 PfSPZ and 4.0x10e5 PfSPZ), followed by 2 groups of adolescents/older children in cohort 2 (each receiving 2.0x10e5 PfSPZ), followed by 1 group of younger children in cohort 3 (receiving 2.0x10e5 PfSPZ). Each group will be composed of 15 participants, 10 to receive PfSPZ-LARC2 Vaccine, and 5 to receive normal saline (NS) placebo, with randomized, blinded, 2:1 allocation to vaccine and placebo in each group. Each group will begin with a pilot group of 2 vaccinees and 1 placebo recipient three or more days before the rest of the cohort initiates, as a safety precaution. In the two cohorts with two groups, the pilot group for the second group will be initiated at least 3 days after the pilot group for the first group. A Safety Monitoring Committee (SMC) will review safety and tolerability data before proceeding to the next cohort.

Each group except group 1 (2.0x10e5 PfSPZ adult group) will receive only a single dose. This is because the risk of breakthrough is thought to be greatest after a first exposure; thereafter, the vaccine-induced immunity from the first dose reduces the risk of breakthrough after subsequent doses . Administering a single "highest-risk-of-breakthrough" first dose in all four age groups allows follow-up without the complexity of intervening second and third immunizations. However, it is theoretically possible (without any supporting evidence) that the biology associated with repeated dosing of LARC2 parasites could be different from this expectation. For this reason, group 1 will be administered second and third doses of 2.0x10e5 PfSPZ, each dose with 28 days of follow-up. It is noted that in the first GA2 trial in Leiden, 9 participants were immunized by mosquito bite three times at monthly intervals and there was no breakthrough after any of the doses. Including 3 doses in group 1 will additionally allow measurement of the immunogenicity of a standard 3-dose regimen for this vaccine (doses on Days 1, 29 and 57) in a malaria-exposed population, allowing comparison with a planned trial in Seattle, where malaria-naive adults will receive the same 3-dose regimen.

Cohort 1:

Group 1 (20-50-year-olds): 15 participants receive 3 injections of 2.0x10e5 PfSPZ or NS (days 1, 29 and 57).

Group 2 (20-50-year-olds): 15 participants receive 1 injection of 4.0x10e5 PfSPZ or NS .

Cohort 2 Group 3 (11-19-year-olds): 15 participants receive 1 injection of 2.0x10e5 PfSPZ or NS.

Group 4 (6-10-year-olds): 15 participants receive 1 injection of 2.0x10e5 PfSPZ or NS.

Cohort 3 Group 5 (1-5-year-olds): 15 participants receive 1 injection of 2.0x10e5 PfSPZ or NS.

Total sample size: 15 x 5 groups = 75 participants, 50 receiving vaccine and 15 placebo.

Two SMC meetings will be scheduled to review safety and tolerability data collected over 28 days in cohorts 1 and 2, respectively. If there are no vaccine strain breakthrough infections in the two cohort 1 groups during 28 days of follow-up after the first dose, and if the vaccine is safe and well-tolerated as revealed by solicited adverse events, unsolicited adverse events, and laboratory abnormalities, the SMC will be asked to recommend proceeding to the next cohort (cohort 2). If there are vaccine strain breakthroughs, the trial will be halted pending review by the SMC, IRBs and regulatory agencies. In like fashion, the SMC will meet a 2nd time to review 28 days of follow-up from cohort 2 and will provide a recommendation regarding the initiation of cohort 3.

To monitor for breakthrough infections following immunization, participants will be followed for 28 days after each immunization for signs and symptoms of malaria by daily recording of solicited and unsolicited adverse events. The likelihood that a given density of parasitemia will be symptomatic is affected by naturally acquired immunity (NAI), which develops gradually during childhood in endemic areas following repeated Pf infection. NAI includes both anti-parasite immunity, which results in lower parasite densities in the blood, and anti-clinical manifestations immunity, which results in reduced signs and symptoms of malaria for a given density of parasitemia. Pre-school malaria-exposed children have minimal NAI and experience the signs and symptoms of malaria at lower parasite densities (e.g., <100 parasites/uL) compared to malaria-exposed adults, who generally limit the density of parasitemia through NAI and may not experience clinical illness unless parasite density exceeds 100-200 parasites/uL. Older children are intermediate in their level of NAI.

Monitoring will also be done by scheduled thick blood smears (TBS), with a frequency based on the following principles: (1) follow-up should be more frequent for cohort 1 (groups 1 and 2), which is planned as first-in-humans; once it is demonstrated that there are no breakthroughs in the first cohort, which includes 10 adults receiving 2.0x10e5 PfSPZ and 10 adults 4.0x10e5 PfSPZ (to augment the risk of breakthrough), the frequency of TBS sampling can be reduced in subsequent cohorts ; (2) blood drawing should be minimized in children to reduce pain and improve compliance, following both Burkinabe and international standards , noting that this diminished TBS frequency is compensated by the fact that parasitemia will clinically manifest at lower parasite densities in children with less NAI than adults, and any symptoms referable to malaria will result in an immediate performance of TBS; (3) to assure safety, it is important that we achieve follow-up in all children; based on Burkinabe experience, parents may withdraw their children from the trial if there are daily needle sticks as planned for the adult cohort, and it is recommended that frequency not exceed every other day to assure compliance.

Based on these considerations, there are different follow-up TBS schedules for adult and pediatric groups. In the adults (groups 1 and 2, first-in-humans), TBS to monitor for Pf blood stage infections will be performed daily from day +6 to day +20 and then every two days until day +28, at which time terminal antimalarial treatment will be administered as a safety measure to group 2 , with a follow-up TBS on day +30 to confirm negativity after 48 hours of treatment (group 1 will receive terminal treatment day +28 after the third dose - see below). Assuming that there are no breakthrough infections in groups 1 and 2 during the first 28 days of follow-up, meaning that the "pre-test probability" of breakthrough infections in the pediatric groups is reduced, and in conformity with research guidelines to minimize the frequency of blood draws in children and to strengthen compliance, the frequency of TBS to detect parasitemia will be reduced in the pediatric age groups to every other day from day +6 to +18, then on days +21, +24 and +28, with terminal treatment initiated on day +28 and a follow-up TBS on day +30 to confirm negativity after 48 hours of treatment. This reduces the number of needle sticks (venipuncture or finger stick) for TBS during the first 30 days from 20 in adults to 11 in children. This is felt to be the maximum number of blood draws with which the pediatric population and their parents/guardians will comply.

As stated earlier, first immunizations induce substantial immunity to Pf malaria. Therefore, TBS follow-up for group 1 after day +28 (the day of the second immunization) will be weekly (+35, +42, +49, +56, +63, +70, +77, and +84 ), with terminal treatment initiated on day +84 and a follow-up TBS on day +86 to confirm negativity after 48 hours of treatment.

Daily monitoring for adverse events by participants, their parent or guardian, and/or clinical staff will take place during the entire 28-day primary follow-up period after the first dose in each group. Participants/parents/guardians will receive strict instructions to notify the clinical staff at any time (day or night) if symptoms develop. For participants (or parents) with phones, there will be daily contact by phone from the clinical staff to ask about symptoms on all days during the first 28 days of follow-up when there is no scheduled clinic visit. If phone contact is not possible, there will be daily home visits by clinical staff when there is no scheduled clinic visit. This close follow-up is the overriding safety feature for all participants. Severe malaria cannot develop in the absence of typical malaria symptoms. In adults with NAI, typical malaria symptoms are consistently experienced at densities above approximately 500 parasites/uL, which is 2 orders of magnitude below the most conservative definition of severe malaria based on parasitemia level (1% parasitemia, which is approximately 50,000 parasites/uL ).

In all age groups, any symptoms consistent with malaria will be immediately investigated clinically, including by TBS, which will be repeated at least daily if the initial TBS is negative and symptoms are grade 1 or 2 in severity, or every 8 to 12 hours if initial TBS is negative and symptoms are grade 3 in severity. Malaria signs and symptoms include fever (axillary temperature in > 37.5°C [>99.5°F]), subjective fever, headache, dizziness, malaise, fatigue, chills, rigors, sweats, myalgia, arthralgia, nausea, vomiting, diarrhea, abdominal pain, cough and chest pain. For pre-verbal children, signs and symptoms will be fever, subjective fever, irritability/fussiness, drowsiness and loss of appetite.

Any density of parasitemia identified by TBS will be considered indicative of malaria infection and will be treated after a sample is obtained to allow genomic analysis of the parasite (to determine if it is vaccine strain or wild-type Pf infection ).

Serious adverse events (SAEs) will be monitored throughout the trial. Laboratory tests (white blood count, neutrophil count, lymphocyte count, hemoglobin, platelets, creatinine, alanine aminotransferase, aspartate aminotransferase) will be done at screening, the day of immunization, and 6 and 28 days after immunization for groups 2, 3, 4 and 5. For group 1, laboratory tests will be done at screening, the day of first immunization, 6 days after the first immunization, the day of second immunization, 7 days after the second immunization, the day of third immunization and 7 and 28 days after the third immunization.

Three and six months (12 and 24 weeks) after the final immunization in each group, there will be follow-up visits to review the participant's health since terminal antimalarial treatment. Because all participants receive terminal treatment prior to this follow-up period, the risk of vaccine-strain induced malaria during this period is low. However, it is theoretically possible that there could be delayed release of parasites from the liver, which is the reason for ongoing follow-up. The drugs used for terminal treatment are primarily active against asexual blood stages and may not kill liver stages. The three doses administered to group 1 (the standard full series) will allow further investigation of LARC2 parasite biology and risk of breakthrough during this added follow-up period. Participants (or their parents / guardians) will be strictly instructed to contact clinical staff for signs or symptoms of malaria during the post terminal treatment period.

Definition of blood stage parasitemia during the immunization phase: Any positive TBS showing normal appearing parasites confirmed by a second reader (with a third reader used to resolve disagreements between the first two). TBS will generally be made from finger-prick blood, but venipuncture can be used if preferred by the participant or if it needs to be done anyway for other tests. TBS will be made according to Sanaria's SOP which provides for quantification of parasite density. TBS will be read in real-time as collected, prioritizing the reading of TBS from symptomatic participants.

If the TBS turns positive during follow-up: If a participant develops parasitemia, they will be treated as soon as parasitemia is identified even if asymptomatic. Treatment will be by DOT (directly observed treatment ). A blood sample adequate for genetic analysis and culture will be obtained by venipuncture prior to treatment. The drugs for treatment will be dihydroartemisinin-piperaquine (DHA-P) with artemether-lumefantrine (AL) as back-up. In addition, a single low dose of primaquine (PQ) will be administered to kill any gametocytes and prevent transmission. Both DHA-P (or AL) and PQ treatments will be appropriately adjusted for body weight. G6PD testing is not required for a single administration of primaquine in this population (0.25 mg/kg).

Given the high likelihood that PfSPZ-LARC2 vaccine is fully attenuated, it is expected that any parasitemias detected in research participants will be caused by naturally acquired infections, as the study will be performed in a malaria endemic area where Pf transmission can occur year-round, even though rates are significantly less in the dry season. However, in order to demonstrate definitively that any parasitemias are derived from wild-type parasites, genetic analyses will be performed on all parasitemias developing during 28 days of follow-up in cohort 1 (groups 1 and 2) before progressing to cohort 2 and during 28 days of follow-up in cohort 2 before progressing to cohort 3 (any parasitemias developing in cohort 1, group 1, from 28 days post first immunization to terminal treatment will be included in this second set of parasitemias).

The prompt genetic assessment will be done using an assay that is similar to that used as an identity test to release the master cell bank and individual lots of PfSPZ-LARC2 Vaccine, although the conditions of the assay are modified for use on whole blood with potentially low density parasitemia. If the test is negative for the genetically engineered parasites, it will indicate that the infection was naturally acquired, and the trial will continue. If the parasite is vaccine strain, the trial will be halted and the SMC, the IRBs (US and Burkina Faso) and the regulatory authorities (US and Burkina Faso) will be informed.

In contrast to the immunization phase, which will be completed during the dry season, the six months of follow-up post terminal treatment will extend into the rainy season. It is therefore anticipated that many if not most participants will acquire naturally transmitted malaria. Blood samples from these infections will be collected for possible future analyses (optional, exploratory endpoint).

Clearance of parasitemia prior to immunization: Because the study is being done in malaria-exposed individuals, some of whom may have chronic parasitemia, it will be essential to clear any existing parasitemia prior to immunization. Otherwise, pre-existing parasitemia could recrudesce during follow-up. As a recrudescing wild-type parasitemia will be indistinguishable clinically or by TBS from breakthrough vaccine strain parasitemia, it will needlessly complicate follow-up.

Clearance will be administered to all participants because it is not possible to determine which participants have latent infection, even if the most sensitive PCR is used. Clearance will be started two weeks before immunization using a three-day treatment course of artemether / lumefantrine (AL) with dosing adjusted for body weight. It will be administered by study staff using DOT. This is one of two artemisinin combination therapies (ACTs) used for treating malaria in Burkina Faso. This particular ACT is selected based on the relatively short half-life of the longer-acting lumefantrine compared to piperaquine, the longer-acting drug of the other ACT used in Burkina Faso, dihydroartemisinin / piperaquine (DHA-P) . A short half-life is needed: (1) to prevent any potential impact on the PfSPZ in the vaccine and their development as liver stages (although even relatively high levels of lumefantrine should not affect liver stages - it acts only against blood stages) and (2) to not interfere with the detection of any breakthrough parasitemias post immunization. Initiating the three-day course on the 14th day prior to immunization and completing the three-day course by the 12th day prior to immunization will assure the passage of at least two half-lives of lumefantrine before immunization and at least three (and more often four or five) half-lives before any breakthrough parasites could appear in the blood, which is six days after immunization.

Terminal treatment four weeks after immunization: As described above, all individuals will be treated 28 days after their first (groups 2, 3, 4, 5) or third (group 1) immunization. DHA-P or AL will be used, as there is no concern about drug half-lives in this case, and both these ACTs are nationally recommended malaria treatments in Burkina Faso.

Treatment of diagnosed parasitemia: The same two ACTs will be used for any parasitemias appearing during the trial.

Seasonal malaria chemoprophylaxis in group 5: One- to five-year-old children in Burkina Faso are placed on seasonal malaria chemoprophylaxis with sulfadoxine/pyrimethamine (SP) during the rainy season, per national guidelines, generally beginning in the month of July at the study site. This will need to be timed so that SP is not administered during the period starting 8 weeks before immunization extending to 4 weeks after immunization in group 5, as SP will interfere with the ability to detect breakthrough infection. The clinical team will ask permission to defer SP administration accordingly. Starting at the time of clearance prior to immunization through to the time of terminal treatment 28 days post immunization, the participants will be monitored daily for signs and symptoms of malaria. If signs or symptoms are present, a TBS will be performed and the participant treated. Thus, there should be no risk to the participant if SP is deferred.

Long-term Follow-up: Participants (or their parents) will be scheduled for in-clinic visits 3 months and 6 months (12 and 24 weeks) after the last immunization to obtain follow-up, to remind them to contact clinical staff for any illness and to record any unrecorded episodes of clinical malaria or SAEs. Clinical malaria that is not identified by the study team in real time during this secondary, post-terminal treatment follow-up period and is reported historically by parents, guardians or participants will be defined as a positive diagnostic test (TBS or rapid diagnostic test) plus fever (as defined previously) plus symptoms consistent with malaria.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males and females, based on clinical and laboratory findings
2. From the age 1 to 50 years
3. Adults with a Body Mass Index (BMI) 18 to 30 Kg/m2; or adolescents, and children with Z-score of the selected indicator ([weight-for-height], [(height and BMI) for age]) category within ±2SD.
4. Residence in the study area for the duration of the study.
5. Agreement to release medical information and to inform the study doctor concerning contraindications for participation in the study
6. Willingness to be attended to by a study clinician and take all necessary medications prescribed during study period
7. Agreement to provide contact information of a third party household member or close friend to study team
8. Agreement not to participate in another clinical trial during the study period
9. Agreement not to donate blood during the study period (until final clearance is completed)
10. Able and willing to complete the study visit schedule over the study follow up period.
11. Willingness to undergo HIV, hepatitis B (HBV), hepatitis C (HCV), and sickle cell anemia tests
12. Volunteer participant (subjects 21 years of age and older) or the parent / guardian signing the informed consent (for subjects <21 years of age) is able to demonstrate their understanding of the study by responding correctly to 9 out of 10 true/false statements (in a maximum of two attempts for those who failed to respond correctly to all true/false statements in the first attempt)
13. Signed written informed consent, in accordance with local practice, provided by adult volunteers, parents or legal representatives and relevant assent for children participants as applicable
14. Has not been treated with any antimalarial medication for at least two weeks prior to the initial clearance treatment.
15. Female volunteers aged 12 years and above must be non-pregnant (as demonstrated by a negative urine pregnancy test), and provide consent / assent of their willingness to take protocol-defined measures not to become pregnant during the study and safety follow-up period. Acceptable measures to not become pregnant include oral or implanted contraceptives, IUD, female condom, diaphragm with spermicide, cervical cap, abstinence, use of a condom by the sexual partner or sterile sexual partner during the entire study. Women with a history of surgical or chemical sterilization (e.g., tubal ligation, hysterectomy, other) must provide written documentation of the procedure from a health care provider.
16. One additional inclusion criterion is demonstration of the ability to complete pre-vaccination drug clearance without significant untoward effects.

Exclusion Criteria:

1. Unable to provide informed consent including inability to pass the test of understanding.
2. Receipt of a malaria vaccine in a prior clinical trial.
3. History of a splenectomy or sickle cell disease.
4. History of a neurologic disorder (including non-febrile seizures or complex febrile seizures) or formal history of migraine headache.
5. Current use of systemic immunosuppressant pharmacotherapy.
6. Receipt of a live vaccine within 4 weeks of first immunization or of 3 or more non-live vaccines within 2 weeks of first immunization.
7. Women who are breast-feeding, pregnant or planning to become pregnant during the study period.
8. Known allergy to atovaquone-proguanil (AP), dihydroartemisinin-piperaquine (DHA-P), artemether-lumefantrine (AL), or any component of the investigational products.
9. History of anaphylaxis or other life-threatening reaction to a vaccine.
10. Participation in any study involving investigational vaccine or drug within 4 weeks prior to enrollment that in the estimation of the site PI might adversely affect the individual's safety or the quality of data to be collected.
11. Evidence of increased cardiovascular disease risk; defined as >10% five-year risk by non-laboratory method (Gaziano, 2008).
12. Plan to participate in another investigational vaccine/drug research during the study.
13. Plan for major surgery between enrollment until last study visit.
14. Use or planned use of any drug with anti-malarial activity that would precede or coincide with vaccination through to 28 days after the last dose of vaccine.
15. Anticipated use of medications known to cause drug interactions with DHAP (antiarrhythmics, neuroleptics, macrolide antibiotics, fluoroquinolones, imidazole and triazole antifungal agents, quinine, halofantrine, pentamidine and saquinavir, certain non-sedating antihistamines, all of which can affect QT intervals - see Section2.2.1.3) or AL (the same list of drugs affecting QT intervals plus rifampin, carbamazepine, phenytoin, St. John's wort and antiretroviral drugs).
16. Positive HIV, HBsAg or HCV serology.
17. History of or evidence for other chronic disease conditions including cancer, diabetes, renal failure, hypertension, tuberculosis, etc.
18. History of arrythmias or cardiac disease, or an abnormal electrocardiogram, defined as one showing prolonged QT interval, pathologic Q waves and significant ST-T wave changes; left ventricular hypertrophy; any non-sinus rhythm including isolated premature ventricular contractions, but excluding isolated premature atrial contractions; right or left bundle branch block; or advanced (secondary or tertiary) A-V heart block; or other clinically significant abnormalities on the electrocardiogram.
19. Any clinically significant deviation from the normal range in biochemistry or hematology tests measured at screening and not resolving (grade 1 abnormalities are allowed).
20. Any medical, psychiatric, social, behavioral or occupational condition or situation (including active alcohol or drug abuse affecting social function) that, in the judgment of the site PI, impairs the participant's ability to give informed consent, increases the risk to the participant of participation in the study, affects the ability of the participant to participate fully in the study, or might negatively impact the quality, consistency, integrity or interpretation of data derived from their participation in the study.
21. One additional exclusion criterion is inability to take a course of malaria treatment prior to receipt of investigational product.

Ages: 1 Year to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-03-04 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Assess safety, namely adequacy of attenuation, of PfSPZ-LARC2 Vaccine by measuring number of trial participants with presence of breakthrough blood stage infection | First 28 days after immunization with PfSPZ-LARC2 Vaccine
  Number of trial participants with presence of breakthrough blood stage infection during the first 28 days after immunization shown to be the vaccine strain.
  Participants will be followed for parasitemia by thick blood smear (TBS) after immunization. TBS to monitor for Pf blood stage infections will be performed every two days from Day 7 (day +6) to Day 19 (day +18) and then on Days 21, 24 and 29 (days +20, +23 and +28) .
Assess the safety of PfSPZ-LARC2 administration by measuring incidence of related grade 3 solicited and unsolicited adverse events (AEs) in the 28 days after PfSPZ-LARC2 Vaccine administration | First 28 days after immunization with PfSPZ-LARC2 Vaccine
  Participants will be followed for solicited and unsolicited adverse events 28 days after immunization. Incidence of possibly related, probably related or definitely related (a) grade 3 solicited adverse events (AEs) in the 28 days after PfSPZ-LARC2 Vaccine administration; and (b) grade 3 unsolicited AEs in the 28 days after PfSPZ-LARC2 Vaccine administration will be measured.
Assess the safety of PfSPZ-LARC2 administration by measuring incidence of related grade 3 abnormal laboratory values one week after PfSPZ-LARC2 Vaccine administration | 7 days after immunization with PfSPZ-LARC2 Vaccine
  Incidence of possibly related, probably related or definitely related grade 3 abnormal laboratory values one week after PfSPZ-LARC2 Vaccine administration;
Assess the safety of PfSPZ-LARC2 administration by measuring incidence of related serious adverse events (SAEs) throughout the study period | Entire study period (approximately 6 months)
  Incidence of possibly related, probably related or definitely related serious adverse events (SAEs) throughout the study period.

SECONDARY OUTCOMES:
To further assess safety following vaccination by measuring incidence of mild to moderate solicited and unsolicited AEs in the 28 days after injection of PfSPZ-LARC2 Vaccine | First 28 days following immunization with PfSPZ-LARC2 Vaccine
  Incidence of mild to moderate (a) solicited adverse events (AEs) in the 28 days after injection of PfSPZ-LARC2 Vaccine; and (b) unsolicited AEs in the 28 days after injection of PfSPZ-LARC2 Vaccine .
To further assess safety following vaccination by measuring incidence of mild to moderate abnormal laboratory values one week after injection of PfSPZ-LARC2 Vaccine | 7 days after immunization with PfSPZ-LARC2 Vaccine
  Incidence of mild to moderate abnormal laboratory values one week after injection of PfSPZ-LARC2 Vaccine.
To identify immune responses following vaccination and their association with age and sex by measuring Anti-P. falciparum circumsporozoite protein antibody levels two weeks after PfSPZ-LARC2 Vaccine administration. | 14 days after immunization with PfSPZ-LARC2 Vaccine
  Anti-P. falciparum circum-sporozoite protein antibody levels measured by ELISA two weeks after PfSPZ-LARC2 Vaccine administration.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas L Dr. Thomas L. Richie, MD PhD, Study Director — Sanaria Inc.
Locations (1):
- Groupe de Recherche Action en Santé (GRAS) / Unité de Recherche Clinique de Sabou, Ouagadougou, Burkina Faso